CLINICAL TRIAL: NCT05457296
Title: Saliva Cortisol Measurement for the Assessment of Hydrocortisone Replacement Therapy in Secondary Adrenal Insufficiency Patients
Brief Title: Salivary Cortisol Measurement in Corticotrope Deficiency Substitution With Hydrocortisone.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Melika Chihaoui, professor, University Tunis El Manar
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 101
Record Dates: First submitted 2021-03-03; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Adrenal Insufficiency
Keywords: Adrenal Insufficiency; hydrocortisone; salivary cortisol; pharmacokinetic
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Hydrocortisone; Capsules

STUDY DESIGN:
Intervention Model Description: prospective case control and randomized crossover clinical trial
Who Masked: Participant, Care Provider
Masking Description: healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- capsule hydrocortisone intake in patients with corticotrope deficiency (Experimental): Hydrocortisone taken in capsule form (15mg), one intake/ one day test.
  Interventions: Drug: Hydrocortisone (capsule)
- tablet hydrocortisone intake in patients with corticotrope deficiency (Active Comparator): Hydrocortisone taken in tablet form (15mg), one intake/ one day test.
  Interventions: Drug: Hydrocortisone (capsule)
- healthy controls (No Intervention): healthy non treated controls, one day test.

INTERVENTIONS:
Drug: Hydrocortisone (capsule) — salivary cortisol measurement at baseline and at one, two, and four hours after hydrocortisone intake.
  Arms: capsule hydrocortisone intake in patients with corticotrope deficiency; tablet hydrocortisone intake in patients with corticotrope deficiency

SUMMARY:
Patients with adrenal insufficiency are most often overdosed with hydrocortisone. To date, there is no reliable marker that can reflect the quality of hydrocortisone substitution. Salivary cortisol is a good reflection of free plasmatic cortisol. However, salivary contamination with the oral intake of hydrocortisone has been described.

The aims of the study are to:

* evaluate the frequency of salivary contamination by hydrocortisone taken in tablet form and determine its risk factors.
* evaluate the quality of hydrocortisone substitution in patients with corticotrope deficiency.

DETAILED DESCRIPTION:
Patients with adrenal insufficiency are most often overdosed with hydrocortisone, as evidenced by the higher frequency of metabolic disorders, osteoporosis and cardiovascular mortality in these subjects compared to healthy subjects. To date, there is no reliable marker that can reflect the quality of hydrocortisone substitution. Salivary cortisol is a good reflection of free plasmatic cortisol. However, salivary contamination with the oral intake of hydrocortisone has been described.

The aims of the study are to:

* evaluate the frequency of salivary contamination by hydrocortisone taken in tablet form and determine its risk factors.
* evaluate the quality of hydrocortisone substitution in patients with corticotrope deficiency.

It is a cross over clinical trial with three arms: patients taking tablets of hydrocortisone, patients taking capsules of hydrocortisone, and healthy control subjects undergoing one day test. Salivary cortisol is measured before, at one, two and four hours after hydrocortisone intake.

ELIGIBILITY:
Inclusion Criteria:

-patients with corticotrope deficiency treated with hydrocortisone for at least one year.

Exclusion Criteria:

* alcoholism,
* morbid obesity,
* long standing or uncontrolled diabetes mellitus,
* uncontrolled hypothyroidism,
* depression,
* chronic or acute inflammatory or infectious disease,
* neoplasia,
* renal or hepatic disease,
* malabsorption,
* pregnant or breast-feeding women,
* treatment with corticosteroids other than hydrocortisone, enzyme inducers or oestrogens.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Oral contamination of salivary cortisol measurement with hydrocortisone taken in tablet form. | during the four hours test
  very high salivary cortisol levels after the intake of hydrocortisone in tablet form as compared with capsule form.

SECONDARY OUTCOMES:
Evaluation of the quality of the substitution of corticotrope deficiency with hydrocortisone using salivary cortisol measurement | salivary cortisol levels during the four hours test
  patients under-treated, over-treated or well treated (comparison of salivary cortisol levels with those of healthy controls)

CONTACTS AND LOCATIONS:
Overall Officials: Meriem Kallel, professor, Study Chair — Research committee of the university hospital La Rabta
Locations (2):
- Tunisia (2):
  - university hospital La Rabta, Tunis
  - University hospital La Rabta, Tunis

IPD SHARING:
Plan to Share IPD: No